CLINICAL TRIAL: NCT00181064
Title: Use of the Atkins Diet for Adolescents With Chronic Daily Headache.
Brief Title: Atkins Diet for Difficult-to-Control Headaches in Teenagers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Eric Kossoff, Johns Hopkins University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-08-10-04
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-06

CONDITIONS: Chronic Daily Headache
Keywords: headache; Atkins; ketosis; intractable
MeSH Terms: conditions — Headache Disorders; Headache; Ketosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Modified Atkins diet — 15 grams of carbohydrates per day - high fat diet

SUMMARY:
This is a 3-month pilot study of 10 adolescents with chronic daily headache. Teens will be placed on a modified Atkins diet and followed with 2 subsequent visits to assess for headache improvement.

DETAILED DESCRIPTION:
Patients are placed on the diet and followed with various measures for 3 months. If the diet is helpful it is continued. Patients are still being enrolled as of 9/6/06.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12-19
* Minimum 15 headaches/month for at least 3 months
* Tried 2 preventative medications previously

Exclusion Criteria:

* Prior use of the Atkins diet for more than 1 week
* Pregnancy
* Significant heart or kidney disease
* Dangerously underweight
* Using acute pain medications more than 11 days in the past month
* Medications being changed

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2005-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Headaches | 3 months

SECONDARY OUTCOMES:
Ketosis | 3 months
Diet duration | as long as tolerated
Quality of life (PedsMIDAS) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric H Kossoff, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Strahlman RS. Can ketosis help migraine sufferers? A case report. Headache. 2006 Jan;46(1):182. doi: 10.1111/j.1526-4610.2006.00321_5.x. No abstract available. PMID 16412174